CLINICAL TRIAL: NCT04319770
Title: Effectiveness of Hyaluronic Acid Versus Enamel Matrix Derivatives in the Regeneration of Infrabony Defects. A Randomized Controlled Clinical Trial
Brief Title: Effectiveness of Hyaluronic Acid in the Regeneration of Infrabony Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea Pilloni MD DDS MS, Chairman Section of Periodontics Director of Master Program in Periodontics, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ref. 3816 - Prot. 2705/15
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Intrabony Periodontal Defect

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- periodontal regenerative surgery + EMD (control) (Active Comparator): periodontal regenerative surgery with enamel matrix derivative
  Interventions: Device: enamel matrix derivative (EMD)
- periodontal regenerative surgery + HA (test) (Experimental): periodontal regenerative surgery with hyaluronic acid
  Interventions: Device: hyaluronic acid (HA)

INTERVENTIONS:
Device: enamel matrix derivative (EMD) — periodontal regenerative surgery with enamel matrix derivative (EMD) (control)
  Arms: periodontal regenerative surgery + EMD (control)
Device: hyaluronic acid (HA) — periodontal regenerative surgery with hyaluronic acid (HA) (test)
  Arms: periodontal regenerative surgery + HA (test)

SUMMARY:
The purpose of this randomized controlled clinical trial (RCT) is to determine the efficacy hyaluronic acid (HA) versus enamel matrix derivatives (EMD) in the treatment of infrabony periodontal defects.

DETAILED DESCRIPTION:
Intrabony defects associated with periodontal pockets represent a risk factor for periodontitis progression and additional loss of attachment if left untreated.

Over the years, several strategies have been implemented for their surgically reconstruction with the aim of pocket reduction and clinical attachment level gain.

Grafting of intrabony periodontal defects has been used extensively over the years incorporating various materials, including autogenic bone, demineralized allogenic bone, xenogenic and alloplastic materials. Controlled clinical studies have shown a significantly higher gain of clinical attachment and radiographic bone gain in intra-bony periodontal defects treated with open flap debridement combined with EMD when compared with open flap debridement alone.

Hyaluronic acid (HAc) is a naturally occurring linear polysaccharide of the extracellular matrix of connective tissue, synovial fluid, and other tissues. It possesses various physiological and structural functions, which include cellular and extracellular interactions, interactions with growth factors and regulation of the osmotic pressure, and tissue lubrication. All these functions help in maintaining the structural and homeostatic integrity of the tissue.

In the field of dentistry, in vitro and animal studies have demonstrated that hyaluronic acid prevents oxygen free-radical damage to granulation tissue, stimulates the clot formation , induces angiogenesis and does not interfere in the calcification nodule during bone formation.

A randomized controlled trial evaluated the effect of local application of 0.8% Hyaluronan gel in conjunction with periodontal surgery. After initial non-surgical periodontal therapy and re-evaluation, defects were randomly assigned to be treated with modified Widman flap surgery in conjunction with either 0.8% Hyaluronan gel (test) or placebo gel (control) application. Statistically, significant differences were noted for Clinical Attachment Level and gingival recession, (P < 0.05) in favor of the test sites. But non-significant results were found regarding PD, BOP and PI values (P > 0.05).

At the present time no comparative data are available about the use of HA versus EMD in treatment of infrabony defects. Therefore the aim of this study will be evaluated the effectiveness of hyaluronic acid versus enamel matrix derivatives alone in the regeneration of infrabony defects.

ELIGIBILITY:
Inclusion Criteria:

Patient related:

* adults aged 18-65 years with periodontal disease
* sites with infrabony defects and persisting pockets [probing pocket depth (PPD) ≥ 5 mm and bleeding on probing (BOP)] at re-evaluation 6 weeks after non-surgical periodontal therapy
* full-mouth plaque score (FMPS)1 and full-mouth bleeding score (FMBS)2 < 20% before surgery
* at least one radiographically detectable infrabony lesion,3
* good physical health.

Site-specific:

* Interproximal angular defects on single-rooted teeth
* radiographic infrabony component ≥ 3 mm
* PPD ≥ 6 mm and CAL ≥ 7 mm.

Exclusion Criteria:

* relevant medical conditions contraindicating surgical interventions
* pregnancy or lactation
* tobacco smoking
* untreated periodontal conditions
* any condition associated with poor compliance or failure to maintain good oral hygiene
* acute infectious lesions in areas intended for surgery
* teeth with grade 2 or higher mobility
* restorations or carious lesions on root surfaces that are associated with the intrabony defect.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-09-06 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
clinical attachment level (CAL) | baseline, 12, 28 and 24 months
  Changes in CAL between initial and final. Measured in mm

SECONDARY OUTCOMES:
probing pocket depth (PPD) | baseline, 12, 28 and 24 months
  Changes in PPD between initial and final. Measured in mm
gingival recession (GR) | baseline, 12, 28 and 24 months
  Changes in GR between initial and final. Measured in mm

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Pilloni, MD,DDS,MS, Study Director — University of Roma La Sapienza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cortellini P, Pini Prato G, Tonetti MS. Periodontal regeneration of human infrabony defects. I. Clinical measures. J Periodontol. 1993 Apr;64(4):254-60. doi: 10.1902/jop.1993.64.4.254. PMID 8483087
- [Result] Esposito M, Grusovin MG, Papanikolaou N, Coulthard P, Worthington HV. Enamel matrix derivative (Emdogain(R)) for periodontal tissue regeneration in intrabony defects. Cochrane Database Syst Rev. 2009 Oct 7;2009(4):CD003875. doi: 10.1002/14651858.CD003875.pub3. PMID 19821315
- [Result] Cortellini P, Prato GP, Tonetti MS. The modified papilla preservation technique. A new surgical approach for interproximal regenerative procedures. J Periodontol. 1995 Apr;66(4):261-6. doi: 10.1902/jop.1995.66.4.261. PMID 7782979
- [Result] Cortellini P, Prato GP, Tonetti MS. The simplified papilla preservation flap. A novel surgical approach for the management of soft tissues in regenerative procedures. Int J Periodontics Restorative Dent. 1999 Dec;19(6):589-99. PMID 10815597
- [Result] Zhao N, Wang X, Qin L, Guo Z, Li D. Effect of molecular weight and concentration of hyaluronan on cell proliferation and osteogenic differentiation in vitro. Biochem Biophys Res Commun. 2015 Sep 25;465(3):569-74. doi: 10.1016/j.bbrc.2015.08.061. Epub 2015 Aug 15. PMID 26284973
- [Result] Vanden Bogaerde L. Treatment of infrabony periodontal defects with esterified hyaluronic acid: clinical report of 19 consecutive lesions. Int J Periodontics Restorative Dent. 2009 Jun;29(3):315-23. PMID 19537471
- [Result] Fawzy El-Sayed KM, Dahaba MA, Aboul-Ela S, Darhous MS. Local application of hyaluronan gel in conjunction with periodontal surgery: a randomized controlled trial. Clin Oral Investig. 2012 Aug;16(4):1229-36. doi: 10.1007/s00784-011-0630-z. Epub 2011 Oct 20. PMID 22012469